CLINICAL TRIAL: NCT07107295
Title: Investigation of Thoracolumbar Fascia Thickness and Its Relationship With Balance, Trunk Control, Trunk Flexibility, and Functional Independence in Chronic Stroke Patients
Brief Title: Thoracolumbar Fascia Thickness in Chronic Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Büşra Seçkinoğulları Korkusuz, Principal Investigator, Ankara University
Other Study IDs: E-59394181-604.01-114825
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Chronic Stroke Patients
- Control Group: Healthy individuals with similar demographic characteristics

SUMMARY:
The main objective of this study was to examine the thoracolumbar fascia thickness in chronic stroke patients using objective methods and to reveal the relationship of this flexibility with balance, trunk control, trunk flexibility, functional independence and other relevant clinical parameters. Demographic information will be recorded and evaluated. Thoracolumbar fascia thickness will be assessed for individuals in both groups using ultrasonography, trunk flexibility using the Sit-and-Reach test, trunk function using the Trunk Impairment Scale, balance using the Functional Reach Test and the Timed Up and Go test, and functional independence using the Functional Independence Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40 and 70 years old.
* Being diagnosed with a stroke by a neurologist.
* Scoring above 21 on the Montreal Cognitive Assessment Scale.
* Scoring between 0 and 3 on the Modified Rankin Scale.
* Being at least 6 months past the stroke

Exclusion Criteria:

* Inability to communicate verbally
* Individuals with severe visual impairment, neurological disorders in addition to stroke, and/or congestive heart failure
* Patients in whom exercise is not recommended.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients between the ages of 40 and 70 who are receiving routine treatment at a Private University Hospital and healthy individuals with similar demographic characteristics will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Assessment | Baseline
  In this study, ultrasonography will be used to assess the thickness of the thoracolumbar fascia in participants. Participants will be assessed in a comfortable prone position. A physical therapist trained in musculoskeletal ultrasonography will measure the thickness of the thoracolumbar fascia at standard anatomical landmarks. During measurements, care will be taken to ensure the probe is placed perpendicularly and steadily against the muscle tissue, and the images will be optimized and recorded to ensure accurate measurement of muscle thickness. Data obtained will be expressed in millimeters and recorded along with the participants' age, gender, and other demographic information.
Sit-and-Reach Test | Baseline
  This study will be used to assess the flexibility of participants' hamstrings and lumbar extensors. This test is a standardized assessment method that measures how far a person can reach in a seated position with their legs straight, typically using a flexibility box or tape measure. Participants will be asked to sit with their legs straight and lean forward, with their feet resting on the measuring box or wall, without bending their knees. They will be asked to touch their toes as far forward as possible. The farthest point they reach will be recorded in centimeters. The test will be repeated twice, and the best performance will be considered. The resulting values will be used in analyses as an indicator of participants' trunk and lower extremity flexibility levels.
Functional Reach Test | Baseline
  This test is a simple and reliable method for measuring static balance, measuring the maximum distance in centimeters a person can extend their arm forward while standing. The participant is asked to stand parallel to a wall, make a fist with their arm flexed 90 degrees at shoulder height, and reach forward as far as possible without losing their balance or lifting their feet off the ground. The distance between the initial toe position and the maximum reach position is recorded. The test will be repeated three times, and the best performances will be evaluated.
Timed up Go Test | Baseline
  The test assesses functional mobility and balance. The participant rises from a chair, walks 3 meters, turns, walks back to the chair, and sits down. The duration of this activity is recorded with a stopwatch. The test can be performed with the individual's usual assistive devices to ensure safety. Multiple attempts are usually required to ensure optimal performance.
Trunk Impairment Scale | Baseline
  This scale consists of three main sections: static sitting balance, dynamic sitting balance, and trunk coordination. The TIS, which contains 17 items in total, has a maximum score of 23, with higher scores indicating greater trunk control and mobility. The assessment will be conducted by a qualified physiotherapist in accordance with established standard procedures. The results obtained from the scale will be used in statistical analyses as an objective indicator of participants' trunk performance and will be an important data source for determining relationships with other functional parameters.
Functional Independence Measure | Baseline
  The test will be used to assess participants' levels of independence in activities of daily living and their care needs.Each item is scored from 1 (complete dependence) to 7 (complete independence), and the total score ranges from 18 to 126. Higher FIM scores indicate greater functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University; Ayşenur Özcan, MSc, Study Chair — Çankırı Karatekin University; Ali Mert Özcan, MSc, Study Chair — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] Yerli S, Yinanc SB, Yagci G, Erbahceci F, Ozcakar L. Thoracolumbar fascia and chronic low back pain in idiopathic lumbar scoliosis: an ultrasonographic study. Eur Spine J. 2024 Jun;33(6):2469-2475. doi: 10.1007/s00586-024-08266-x. Epub 2024 Apr 23. PMID 38653872